CLINICAL TRIAL: NCT01304381
Title: Integrated Cardiac Care and Palliative Homecare for Patients With Severe Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Association of Local Authorities and Regions (Other)
Responsible Party: Principal Investigator, Margareta Brännström, Senior lecturer, Umeå University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HOPE001
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure; Palliative care; Integrated care
MeSH Terms: conditions — Heart Failure | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated care (Experimental): Multidisciplinary approach and collaboration between specialist palliative and heart failure (HF) caregivers in a shared structured person-centred and identity-promoting homecare
  Interventions: Other: Integrated care
- control (No Intervention): Usual care is performed for the control group

INTERVENTIONS:
Other: Integrated care — Intervention Multidisciplinary approach and collaboration between specialist palliative and heart failure caregivers, in a shared structured person-centred and identity-promoting care during 6 months
  Arms: Integrated care
Other: Integrated care — One group with 31 participants is offered a multidisciplinary approach and collaboration between specialist palliative and heart failure caregivers in a shared structured person-centred care at home. Assessment of need, length of visits and phone calls are planned to be adapted for each patient. After 6 months (+ - two weeks) the patients will be transferred to usual care provider following an established individual care plan.
  Arms: Integrated care

SUMMARY:
Patients with severe heart failure have as many symptoms as many patients with cancer but yet do not have equal access to supportive and palliative care. They have an unpredictable course of illness, which makes difficult to judge when the palliative stage has been reached. The Heart failure and Palliative care Programme is a three-year project in Sweden financed by the Swedish Association of Local Authorities and Regions (SALAR). The overall aim is to develop, implement and evaluate a model that integrates cardiac care and palliative advanced home care for patients with severe chronic heart failure. The primary aim is to study the effects on patients' symptom burden, quality of life and activities of daily living. A randomized controlled clinical study is planned.

Patients (n=62) with a confirmed diagnosis in accordance with the criteria proposed by the European Society of Cardiology and with NYHA III-IV symptoms and at least one of following criteria will be included;

1. At least one episode of worsening heart failure that resolved with injection / infusion of diuretics or the addition of other heart failure treatment in the last 6 months and regarded optimally treated according to the responsible physician.
2. Need for infusions-treatment.
3. Chronic poor quality of life (VAS < 50)
4. Signs of cardiac cachexia (involuntary non-oedematous weight loss ≥ 6% of total body weight within the last 6-12 months)
5. less than one year life expectancy The participants will be randomized to intervention or control group. The intervention consist of a multidisciplinary approach and collaboration between specialist palliative and heart failure (HF) caregivers, in a shared structured person-centred and identity-promoting care at home during six months. Usual care is performed for the control group.

ELIGIBILITY:
Patients with a confirmed diagnosis in accordance with the criteria proposed by the European Society of Cardiology and with NYHA III-IV symptoms. And at least one of following criteria;

1. At least one episode of worsening heart failure that resolved with injection / infusion of diuretics or the addition of other heart failure treatment in the last 6 months and regarded optimally treated according to the responsible physician.
2. Need for infusions-treatment.
3. Chronic poor quality of life (VAS < 50)
4. Signs of cardiac cachexia (involuntary non-oedematous weight loss ≥ 6% of total body weight within the last 6-12 months)
5. less than one year life expectancy.

Exclusion Criteria:

Ineligible are patients:

1. who do not want to participate in the study;
2. with severe communication problems;
3. with severe dementia;
4. with other serious disease in which heart failure is of secondary importance;
5. with other life-threatening illness as the primary diagnosis with expected short survival;
6. when the Primary Care Center which is responsible for patient care is geographically located from more than 30 km radius outside the hospital; and
7. participating in another clinical trial. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
changes from baseline values of symptom scores on the the Edmonton assessment scale (ESAS) after intervention of 4, 12 and 24 weeks | baseline and after 4, 16 and 24 weeks

SECONDARY OUTCOMES:
changes from baseline value of quality of life scores on the EQ-5D and activities in daily life (ADL) after intervention of 4, 12 and 24 weeks | baseline, after 4,16 and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Skellefteå hospital, Skellefteå, Västerbotten County, Sweden

REFERENCES:
- [Background] Brännström M, Brulin C, Norberg A, Boman K, Strandberg G (2005). Being a palliative nurse for persons with severe congestive heart failure in advanced homecare. European Journal of Cardiovascular Nursing, 2005;4 (4):314-323. Brännström M, Ekman I, Norberg A, Boman K, Strandberg G. Living with severe chronic heart failure in palliative advanced home care. European Journal of Cardiovascular Nursing, 2006;5(4):295-302. Brännström M, Ekman I, Boman K, Strandberg G. Being a close relative of a person with severe chronic heart failure in palliative advanced home care - a comfort but also a strain. Scandinavian Journal of Caring Sciences, 2007;21(3):338-344 . Brännström M, Ekman I, Boman K, Strandberg G. Narratives of a man with severe chronic heart failure and his wife in palliative advanced home care over a 4.5-year period. Contemporary Nurse, 2007;27(2):10-22. Brännström M, Björck M, Strandberg G, Wanhainen A. Patients' experiences of being informed about having an abdominal aortic aneurysm - A follow-up case study five years after screening. Journal of Vascular Nursing, 2009;27(3):70-4. Lundman B, Brännström M, Hägglund L, Strandberg G. Fatigue in elderly with chronic heart failure: an under-recognized symptom. Aging Health, 2009;5,(5):619-624. Kristofferzon ML, Johansson I, Brännström M, Arenhall E, Baigi A Brunt D, Fridlund B, Nilsson U, Persson S, Rask M, Wieslander I, Ivarsson B and the SAMMI-study group. Evaluation of a Swedish version of the Watts Sexual Function Questionnaire (WSFQ) in persons with heart disease: A pilot study. European Journal of Cardiovascular Nursing 2010;9(3):168-174 Brännström M, Forssell A, Pettersson B. Physicians' experiences of palliative care for heart failure patients. European Journal of Cardiovascular Nursing, 2011;10(1):64-69.
- [Derived] Talabani N, Angerud KH, Boman K, Brannstrom M. Patients' experiences of person-centred integrated heart failure care and palliative care at home: an interview study. BMJ Support Palliat Care. 2020 Mar;10(1):e9. doi: 10.1136/bmjspcare-2016-001226. Epub 2017 Jul 7. PMID 28689185
- [Derived] Markgren R, Brannstrom M, Lundgren C, Boman K. Impacts of person-centred integrated chronic heart failure and palliative home care on pharmacological heart failure treatment: a substudy of a randomised trial. BMJ Support Palliat Care. 2019 Mar;9(1):e10. doi: 10.1136/bmjspcare-2015-000894. Epub 2016 Jan 20. PMID 26792391
- [Derived] Sahlen KG, Boman K, Brannstrom M. A cost-effectiveness study of person-centered integrated heart failure and palliative home care: Based on a randomized controlled trial. Palliat Med. 2016 Mar;30(3):296-302. doi: 10.1177/0269216315618544. Epub 2015 Nov 24. PMID 26603186
- [Derived] Brannstrom M, Boman K. Effects of person-centred and integrated chronic heart failure and palliative home care. PREFER: a randomized controlled study. Eur J Heart Fail. 2014 Oct;16(10):1142-51. doi: 10.1002/ejhf.151. Epub 2014 Aug 27. PMID 25159126
- [Derived] Brannstrom M, Boman K. A new model for integrated heart failure and palliative advanced homecare--rationale and design of a prospective randomized study. Eur J Cardiovasc Nurs. 2013 Jun;12(3):269-75. doi: 10.1177/1474515112445430. Epub 2012 May 28. PMID 22645405